CLINICAL TRIAL: NCT01216462
Title: First Prospective Observational Registry of the Lazio Regional Network for Acute Coronary Syndromes
Brief Title: Registry of Acute Coronary Syndromes in the Lazio Region of Italy
Acronym: NET-SCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Filippo Neri General Hospital (Other)
Collaborators: Associazione Nazionale Medici Cardiologi Ospedalieri (Other)
Responsible Party: Principal Investigator, Furio Colivicchi, Director, Division of Cardiology, San Filippo Neri General Hospital, Rome, ITALY, San Filippo Neri General Hospital
Other Study IDs: SFN/117/09/AL
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The NET-SCA Registry has been designed to document and evaluate the clinical epidemiology and current management of Acute Coronary Syndromes in the Lazio Region of Italy.

DETAILED DESCRIPTION:
Lazio is a region of central Italy with a resident population of about 5,600,000. The NET-SCA Registry has been designed to document and evaluate the current presentation and clinical management of Acute Coronary Syndromes (ACS) in this specific regional area of Italy. All consecutive patients with ACS admitted to CCU of 15 hospitals of the Lazio Region will be included in the registry.

ELIGIBILITY:
Inclusion Criteria:

* admission to CCU for ACS

Exclusion Criteria:

* ACS due to major extracardiac causes (i.e. traumatic)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with ACS admitted to CCU of 15 hospitals of the Lazio Region of Italy.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Total Mortality | 12 months

SECONDARY OUTCOMES:
Cardiovascular Mortality | 12 months
New admissions of ACS | 12 months
New admissions for heart failure | 12 months
New admissions for coronary revascularization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Furio Colivicchi, MD, Principal Investigator — San Filippo Neri Hospital, Rome, Italy
Locations (8):
- Italy (8):
  - Ospedale "G.B. Grassi", Rome, Italy
  - San Filippo Neri Hospital, Rome, Italy
  - Ospedale "S. Eugenio", Rome, Italy
  - Ospedale "Sandro Pertini", Rome, Italy
  - Policlinico Casilino, Rome, Italy
  - Ospedale "Madre Giuseppina Vannini", Rome, Italy
  - Ospedale FBF "Isola Tiberina", Rome, Italy
  - Ospedale GG Grassi, Ostia Antica, Roma